CLINICAL TRIAL: NCT05629741
Title: A 2-Part First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of CMTX-101, an Anti-DNABII Monoclonal Antibody, in Healthy Subjects (Part 1) and Hospitalized Subjects with Suspected or Confirmed Community-Acquired Bacterial Pneumonia of Moderate Severity (Part 2)
Brief Title: A 2-Part First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of CMTX-101
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped due to slow enrollment. No safety issues were identified. Part 1 (healthy volunteers) fully enrolled; Part 2 (CABP patients) enrolled the first 2 cohorts. Data currently under review. Results will be posted when final.
Sponsor: Clarametyx Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CMTX101-P1-CT001
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Community-acquired Pneumonia; Bacterial Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- CMTX-101 2.5 mg/kg (Experimental): CMTX-101 will be administered as a single IV infusion over 60 minutes.
  Interventions: Drug: CMTX-101
- CMTX-101 5 mg/kg (Experimental): CMTX-101 will be administered as a single IV infusion over 60 minutes.
  Interventions: Drug: CMTX-101
- CMTX-101 15 mg/kg (Experimental): CMTX-101 will be administered as a single IV infusion over 60 minutes.
  Interventions: Drug: CMTX-101
- CMTX-101 30 mg/kg (Experimental): CMTX-101 will be administered as a single IV infusion over 60 minutes.
  Interventions: Drug: CMTX-101
- CMTX-101 0 mg/kg (Placebo Comparator): Placebo will be administered as a single IV infusion over 60 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CMTX-101 — Administered as specified in the treatment arm
  Arms: CMTX-101 15 mg/kg; CMTX-101 2.5 mg/kg; CMTX-101 30 mg/kg; CMTX-101 5 mg/kg
Drug: Placebo — Administered as specified in the treatment arm
  Arms: CMTX-101 0 mg/kg

SUMMARY:
CMTX-101 is a bacterial biofilm disrupting monoclonal antibody being developed as an adjunct therapy with standard of care antibiotics. The goal of this clinical trial is to assess the safety and tolerability of CMTX-101 in healthy volunteers followed by a similar assessment in patients with suspected or confirmed community acquired bacterial pneumonia of moderate severity.

The main questions the study aims to answer are:

* Are single ascending doses of a CMTX-101 intravenous (IV) infusion safe and tolerated
* What is the pharmacokinetic (PK) profile of single-ascending doses CMTX 101
* Do single ascending doses of CMTX 101 induce development of anti-drug antibodies (ADA) and neutralizing antibodies (Nabs)

Exploratory efficacy biomarkers will also be measured in the patient part of the study. Participants will be administered a single IV infusion of CMTX-101 over a 60-minute period; patients will receive the infusion after starting standard of care antibiotics.

ELIGIBILITY:
Inclusion criteria for Part 1 and Part 2

1. Is ≥ 18 years of age at Screening;
2. Is able to provide written informed consent;
3. If a female subject of non-childbearing potential, is either surgically sterile (i.e., has had a hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy at least 26 weeks before Screening) or post-menopausal, defined as spontaneous amenorrhea for at least 2 years, with a follicle-stimulating hormone in the post-menopausal range obtained during Screening;
4. Contraceptive requirements: If a female subject of childbearing potential (i.e., ovulating, pre-menopausal, and not surgically sterile) with a male partner or a male subject with a female partner, must use a medically accepted contraceptive regimen during her/his participation in the study and for 4 months after the last infusion of study drug. Medically accepted contraceptive methods are defined as those with 90% or greater efficacy;

   Acceptable methods of contraception for male subjects include the following:
   1. Condoms with spermicide;
   2. Surgical sterilization of subject (i.e., vasectomy) at least 26 weeks before Screening; or
   3. Sexual abstinence (i.e., refraining from heterosexual intercourse), if the preferred and usual lifestyle of the subject.

      Acceptable methods of contraception for female subjects include the following:
   4. Bilateral tubal ligation, completed at least 12 weeks prior to Screening;
   5. Intrauterine device used for at least 12 weeks prior to Screening;
   6. Hormonal contraception (oral, implant, injection, ring, or patch) for at least 12 weeks prior to Screening;
   7. Diaphragm used in combination with spermicide; or
   8. Sexual abstinence (i.e., refraining from heterosexual intercourse), if the preferred and usual lifestyle of the subject.
5. If a male subject, must agree to abstain from sperm donation through 4 months after infusion of the last dose of study drug;
6. If a female of childbearing potential, must demonstrate a negative serum pregnancy test at Screening and prior to study drug administration;

   Inclusion criteria for Part 1 only (healthy volunteers)
7. Is in general good health, based upon the results of medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG), as judged by the Investigator;
8. Agrees to stay in contact with the site for the duration of the study and provide updated contact information as necessary;
9. Agrees to avoid elective surgery for the duration of the study;

   Inclusion criteria for Part 2 only (subjects with CABP)
10. Has known or suspected CABP requiring hospitalization with the following criteria at any time during the Screening period:

    a. Presents with at least 2 of the following symptoms:

    i. Difficulty breathing; ii. New-onset cough or worsening of baseline cough; iii. Purulent sputum production; or iv. Pleuritic chest pain due to pneumonia.

    b. Has at least 1 of the following vital sign abnormalities:

    i. Fever (oral or tympanic temperature ≥38.3°C [≥100.9°F]) or hypothermia (oral or tympanic temperature <36.0°C [<96.8°F]) within 24 hours of screening: this can be documented by the patient or a health care provider ii. Tachycardia (heart rate >100 bpm); or iii. Tachypnea (respiratory rate >20 breaths per minute).

    c. Has at least 1 of the following signs:

    i. Hypoxemia, defined as an oxygen saturation <92% room air or while receiving supplemental oxygen at the subject's baseline requirement OR a PaO2 <60 mmHg; ii. Clinical evidence of pulmonary consolidation defined as auscultatory and/or percussion findings consistent with pneumonia (e.g., crackles, egophony, dullness); or iii. Leukocytosis, defined as a peripheral white blood cell (WBC) count >10,000/mm3, >15% immature neutrophils (bands) regardless of total WBC count, or leukopenia, defined as a total WBC count <4500 mm3.

    d. Has radiographic evidence of pneumonia within 48 hours before Screening (i.e., infiltrates in a lobar or multi-lobar distribution or diffuse opacities on a chest X-ray or computed tomography scan consistent with bacterial pneumonia); and

    e. Has pneumonia suspected or confirmed of bacterial etiology. Note: The aforementioned symptoms and signs do not have to occur simultaneously at 1 given time point to meet the criterion but must occur during the Screening period.

Exclusion criteria for Part 1 and Part 2

1. Has a history or evidence of systemic autoimmune disease;
2. Has received immunoglobulin or blood products within 120 days prior to Screening;
3. Has a known history or evidence of HIV infection;
4. Has a known history or evidence of chronic hepatitis B defined as persistent hepatitis B surface antigen for >6 months, or has an active hepatitis C virus (HCV) infection, defined as positive HCV RNA; Note: Patients with positive HCV antibodies and negative HCV RNA will be permitted.
5. Has a positive test for drugs of abuse at Screening (both parts) or Day -1 (Part 1);
6. Is participating, plans to participate during the study period, or has participated within the last 30 days prior to Screening in any other investigational study;
7. Has received an investigational drug or live vaccine within 30 days or 5 half-lives of the investigational compound, whichever is longer, prior to Screening;
8. Is currently pregnant or lactating/nursing;
9. Has a history or evidence of an allergic reaction that, in the opinion of the Investigator, may compromise the safety of the subject;
10. Has a known or suspected hypersensitivity to CMTX-101 or its excipients;
11. Has a history or presence of an abnormal 12-lead ECG that, in the opinion of the Investigator, is clinically significant or a QTcF ≥450 milliseconds for males and ≥470 milliseconds for females at Screening (both parts) or Day -1 (Part 1); Note: the exclusion criterion should be evaluated based upon the average of the triplicate 12-lead ECG performed at Screening or Day -1 (Part 1)
12. Has a history or evidence of any other acute or chronic disease that, in the opinion of the Investigator, may interfere with the evaluation of the safety or immunogenicity of the drug or compromise the safety of the subject;

    Exclusion criteria for Part 1 only (healthy volunteers)
13. Has an oral temperature ≥37.5°C (≥99.5°F) at Screening or Day -1;
14. Has an abnormal WBC count, hemoglobin, or platelet count (i.e., >1.5 x upper limit of normal [ULN] or >0.5 x below the lower limit of normal (LLN) per the local laboratory or deemed to be clinically significant per the Investigator) at Screening or Day -1;
15. Has an abnormally elevated alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase (ALP), blood urea nitrogen, or creatinine (i.e., >1.5 x ULN per the local laboratory) at Screening or Day -1;
16. Has an abnormal urinalysis at Screening or Day -1 that, in the opinion of the Investigator, is clinically significant;
17. Is positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) using a rapid antigen test at Day -1;
18. Has received immunosuppressive medications within 45 days prior to Screening;
19. Is unable or unwilling to stop all prescription or over-the-counter medications (other than contraceptive medications) from 14 days prior to dosing until the end of the study;

    Exclusion criteria for Part 2 only (subjects with CABP)
20. Has hospital-acquired bacterial pneumonia, defined as pneumonia developed ≥48 hours after a hospital admission;
21. Requires mechanical ventilation, defined as 1 of the following:

    1. Endotracheal intubation;
    2. Oxygen delivered by high-flow nasal cannula with flow rates >20 L/minute with an FiO2 of ≥0.5; or
    3. Non-invasive positive pressure ventilation.
22. Has hypotension, defined as a systolic blood pressure <90 mmHg;
23. Has known evidence of bone marrow suppression defined as the following:

    1. Leukocytes <3000 cells/µL;
    2. Absolute neutrophil count <1500 cells/µL;
    3. Platelets <100,000/µL; or
    4. Hemoglobin <8 g/dL.
24. Has known liver function test abnormalities defined as the following:

    1. Total bilirubin >1.5 x ULN;
    2. ALT and/or AST >3 x ULN; or
    3. ALP >2.5 x ULN.
25. Has a known estimated glomerular filtration rate <30 mL/min;
26. Has received >24 hours of IV antibiotic administration during the current hospitalization for CABP; Note: Patients who have received IV standard-of-care antibiotics for >24 hours but ≤36 hours during their hospitalization may be considered for enrollment on a case-by-case basis after Medical Monitor and/or Sponsor approval.

    Note: There is no restriction on the duration of outpatient antibiotics that the patient may have received prior to hospitalization;
27. Has a confirmed or suspected pleural empyema (does not include sterile parapneumonic effusion);
28. Has known or suspected meningitis, endocarditis, or osteomyelitis;
29. Has a history of post-obstructive pneumonia;
30. Has suspected or confirmed active primary lung cancer or another malignancy metastatic to the lungs;
31. Has a noninfectious cause of pulmonary infiltrates (i.e., pulmonary embolism, chemical pneumonitis, congestive heart failure, lung cancer, or cystic fibrosis);
32. Has a known or suspected pneumonia of viral etiology, confirmed by a rapid viral diagnostic panel; Note: If a viral respiratory panel has not been collected within the 24 hours prior to Screening, a viral respiratory panel will be administered at Screening to determine eligibility. At a minimum, the panel will evaluate for respiratory syncytial virus, influenza A, influenza B and SARS-CoV-2.
33. Has known severe immunosuppression, including but not limited to receipt of corticosteroid therapy (i.e., ≥20 mg of prednisone/day or equivalent for >4 weeks) within the previous 8 weeks, solid organ or bone marrow transplantation within the previous 12 months, or is currently receiving cytotoxic chemotherapy; or
34. Has a life expectancy of ≤3 months because of any disease or has a medical, psychiatric, occupational, or substance abuse problem that, in the opinion of the Investigator, will make it unlikely that the subject will comply with the Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Number and % of healthy subjects experiencing Adverse Events following ascending doses of a single CMTX-101 IV infusion | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Primary objective of Part 1
Number and % of healthy subjects experiencing Serious Adverse Events following ascending doses of a single CMTX-101 IV infusion | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Primary objective of Part 1
Number and % of healthy subjects experiencing Solicited Adverse Events following ascending doses of a single CMTX-101 IV infusion | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Primary objective of Part 1
Number and % of hospitalized subjects with suspected or confirmed CABP of moderate severity experiencing Adverse Events following dosing of a single CMTX-101 IV infusion | Day 1 to Day 35
  Primary objective of Part 2
Number and % of hospitalized subjects with suspected or confirmed CABP of moderate severity experiencing Serious Adverse Events following dosing of a single CMTX-101 IV infusion | Day 1 to Day 35
  Primary objective of Part 2
Number and % of hospitalized subjects with suspected or confirmed CABP of moderate severity experiencing Solicited Adverse Events following dosing of a single CMTX-101 IV infusion | Day 1 to Day 35
  Primary objective of Part 2

SECONDARY OUTCOMES:
Assess the CMax - Observed maximum plasma concentration determined by ELISA following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the TMax - Time to reach maximum plasma concentration determined by ELISA following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the AUC0-last Area under the concentration time curve following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the AUC0-∞ Area under the concentration time curve from zero to infinite time following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the Terminal phase elimination rate determined by ELISA following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the Terminal elimination half-determined by ELISA following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the Apparent total body clearance (CL/F) determined by ELISA following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the Apparent volume of distribution (Vz/F) determined by ELISA following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Evaluate the immunogenicity of CMTX-101 as measured by anti-drug antibodies (ADAs) determined by electrochemiluminescence assay following ascending doses of a single CMTX-101 IV infusion in healthy subjects | Cohorts 1 and 2: Day 1 to Day 29. Cohorts 3 and 4: Day 1 to Day 100.
  Secondary objective of Part 1
Assess the CMax - Observed maximum plasma concentration determined by ELISA following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the TMax - Time to reach maximum plasma concentration determined by ELISA following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the AUC0-last Area under the concentration time curve following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the AUC0-∞ Area under the concentration time curve from zero to infinite time following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the Terminal phase elimination rate determined by ELISA following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the Terminal elimination half-determined by ELISA following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the Apparent total body clearance (CL/F) determined by ELISA following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Assess the Apparent volume of distribution (Vz/F) determined by ELISA following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2
Evaluate the immunogenicity of CMTX-101 as measured by anti-drug antibodies determined by electrochemiluminescence assay following a single dose of a CMTX-101 IV infusion in hospitalized subjects with suspected or confirmed CABP of moderate severity | Day 1 to Day 35
  Secondary objective of Part 2

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Augusta University Health, Augusta, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - University of Louisville, Louisville, Kentucky
  - Wayne State University, Detroit, Michigan
  - Buffalo VA Medical Center, Buffalo, New York
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Virginia School of Medicine, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No